CLINICAL TRIAL: NCT04186039
Title: Functional Magnetic Resonance Imaging - Blood Oxygenation Level Dependent (MRI-BOLD) of the Feta Lung in Congenital Diaphragmatic and Parietal Malformations
Brief Title: Functional Evaluation of the Fetal Lung by Functional Magnetic Resonance Imaging - Blood Oxygenation Level Dependent (MRI-BOLD), in Congenital Diaphragmatic and Parietal Malformations
Acronym: BOLD FETUS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study manager's decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Filière des Maladies Rares Abdomino-THOraciques : FIMATHO (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP191058; 2019-A02623-54 (Other: ID-RCB Number)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2022-11

CONDITIONS: Congenital Diaphragmatic Hernia; Omphalocele; Gastroschisis
Keywords: Functional magnetic resonance imaging; Blood Oxygen Level Dependent effect; Congenital diaphragmatic hernia; Omphalocele; Gastroschisis; Fetal lung; Respiratory failure
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hernia, Umbilical; Gastroschisis; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Congenital diaphragmatic and parietal malformations (Experimental): Patients with fetal magnetic resonance imaging as part of their usual medical care, for fetal / placental indications of diaphragmatic hernia, omphalocele or gastroschisis.
  Interventions: Diagnostic Test: Functional magnetic resonance imaging - Blood Oxygenation Level Dependent

INTERVENTIONS:
Diagnostic Test: Functional magnetic resonance imaging - Blood Oxygenation Level Dependent — First Functional magnetic resonance imaging - Blood Oxygenation Level Dependent sequence under ambient air.
  Oxygenation of 5 minutes at a rate of 12 l / min. Second Functional magnetic resonance imaging - Blood Oxygenation Level Dependent sequence.

SUMMARY:
The objective is to evaluate the quality of the response to the Blood Oxygen Level Dependent effect in fetuses with diaphragmatic hernias and abdominal wall malformations and to correlate with postnatal respiratory outcome. Pulmonary involvement is a constant in diaphragmatic hernias, it is classic in omphaloceles and especially hepatomphaloceles, and exceptional in laparoschisis. As this is an original exploratory study, no preliminary data are available.

If a correlation is found, the Blood Oxygen Level Dependent effect of the fetal lung may be considered as an early functional marker of postnatal lung function. It can be used in addition to lung-to-head-ratio during prenatal counseling.

The final goal is to be able to detect early in the fetus pulmonary insufficiency to help prenatal counseling and perinatal care.

DETAILED DESCRIPTION:
During the fetal period, there is in the lungs a permanent flow and pressure variations between the "inhaled" amniotic fluid and alveolar secretions, which are essential for pulmonary development. A disruption of this physiological mechanism can induce disorders of the respiratory function, which go from simple delay of maturation to hypoplasia. Respiratory function involves the thoracic muscles (diaphragmatic and intercostal) but also the abdominal muscles, that explains why breathing difficulties are found at birth in neonates with diaphragmatic hernia but also abdominal wall malformations.

This pulmonary involvement highly contributes to the morbidity observed at birth, for which strong prenatal predictive criteria are lacking.

Pulmonary volume measurement by the lung-to-head-ratio is widely used for diaphragmatic hernia has been extended to other congenital malformations, because no other available criteria. The lung-to-head-ratio is a parameter well correlated with survival but insufficiently with morbidity and sequelae.

New functional imaging techniques are in development. Among them, the Blood Oxygen Level Dependent uses hemoglobin as an endogenous contrast agent. It is based on the comparison of a basic status in ambient air with status after oxygenation. It gives a functional evaluation of the organs. But this technique has never been evaluated in the fetal lung yet.

The objective of the study is to evaluate the quality of the response to the Blood Oxygen Level Dependent effect in fetuses with diaphragmatic hernias and abdominal wall malformations and to correlate with postnatal respiratory outcome. It is an original exploratory study and no preliminary data are thus available.

If a correlation is found, the Blood Oxygen Level Dependent effect of the fetal lung may be considered as an early functional marker of postnatal lung function. It could then be used in addition to lung-to-head-ratio during prenatal counseling. The final goal is to be able to detect early in the fetus pulmonary insufficiency to help prenatal counseling and perinatal care.

ELIGIBILITY:
Inclusion Criteria:

* Major patient,
* patient with a simple pregnancy,
* patient between 28 and 33 weeks of amenorrhea,
* patient undergoing fetal MRI as part of their usual care, for fetal / placental indications : diaphragmatic hernia, omphalocele and laparoschisis,
* informed consent signed by the patient and the investigator,
* patient affiliated to a social security scheme (beneficiary or beneficiary).

Exclusion Criteria:

* Patient with one of the usual contraindications for MRI,
* claustrophobic patient,
* patient with an abdominal perimeter> 125 cm,
* patient with multiple-birth pregnancy,
* patient with a pregnancy at the end of a long course of medical assisted procreation,
* patient with chronic respiratory disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Value of the Blood Oxygenation Level Dependent of the fetal lung | 30 months
  Regions of interest (ROI) were manually identified on MRI images, with the largest possible homogenous 2D area. For the lungs, the ROIs were delineated at the maximal chest circumference, delineating the right lung, the left lung.
  Changes in haemoglobin concentration will be evaluated by the variation in transverse R2* signal induced by oxygenation in the delimited ROI.
  The BOLD response will be calculated for each case as the difference between normoxic and hyperoxic period (∆R2*) normalized by normoxic value: ∆R2* = [R2*(norm)-R2*(hyper)] / R2*(norm).
Postnatal respiratory evolution | 30 months
  Duration of mechanical ventilation

SECONDARY OUTCOMES:
Postnatal survival | 30 months
  Survival rate at 30 days after birth
Duration of oxygen dependence | 30 months
  Total days of oxygen requiring
Length of hospitalization | 30 months
  Total days of the neonatal hospitalization before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Naziha KHEN-DUNLOP, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Laurent SALOMON, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No